CLINICAL TRIAL: NCT02560441
Title: A Multicenter Phase II Trial to Evaluate the Safety and Efficacy of IPGDP Regimen Chemotherapy in Patients With Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type
Brief Title: Trial of IPGDP Regimen Chemotherapy in Patients With Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: 307 Hospital of PLA (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Hospital of China Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Hebei Medical University Fourth Hospital (Other); Qilu Hospital of Shandong University (Other); Shandong Cancer Hospital and Institute (Other); Nanfang Hospital, Southern Medical University (Other); Guangdong Provincial People's Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Xuzhou Medical University (Other); Shanxi Province Cancer Hospital (Other); Shanxi Dayi Hospital (Other); Zhangzhou Municipal Hospital of Fujian Province (Other)
Responsible Party: Principal Investigator, Shi Yuankai, vice president, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-LYM-005
Record Dates: First submitted 2015-09-11; First posted 2015-09-25 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chemotherapy followed by radiotherapy (Other): Patients receive 3 cycles of IPGDP (ifosfamide 1.2g/m2 iv on days 3-5; pegaspargase 2000U/m2 im on day 1; gemcitabine 800mg/m2 iv on days 3,8; cisplatin 25 mg/m2 iv on days 3-5; dexamethasone 20mg/m2 iv on days 3-6) chemotherapy followed by radiotherapy.
  Interventions: Other: chemotherapy followed by radiotherapy
- radiotherapy followed by chemotherapy (Other): Patients receive radiotherapy followed by 3 cycles of IPGDP (ifosfamide 1.2g/m2 iv on days 3-5; pegaspargase 2000U/m2 im on day 1; gemcitabine 800mg/m2 iv on days 3,8; cisplatin 25 mg/m2 iv on days 3-5; dexamethasone 20mg/m2 iv on days 3-6) chemotherapy.
  Interventions: Other: radiotherapy followed by chemotherapy
- IPGDP regimen chemotherapy (Other): Patients receive 6 cycles of ifosfamide 1.2g/m2 iv on days 3-5; pegaspargase 2000U/m2 im on day 1; gemcitabine 800mg/m2 iv on days 3,8; cisplatin 25 mg/m2 iv on days 3-5; dexamethasone 20mg/m2 iv on days 3-6. 6 cycles, every 3 weeks one cycle.
  Interventions: Drug: IPGDP regimen chemotherapy

INTERVENTIONS:
Other: chemotherapy followed by radiotherapy
  Arms: chemotherapy followed by radiotherapy
Other: radiotherapy followed by chemotherapy
  Arms: radiotherapy followed by chemotherapy
Drug: IPGDP regimen chemotherapy
  Arms: IPGDP regimen chemotherapy

SUMMARY:
The first Part: recruiting untreated ENKL patients with extensive stage I or limited stage II disease (only referring to patients with the invasion of Waldeyer's ring and cervical lymph nodes) . Patients are randomly divided into two arms, IPGDP regimen chemotherapy followed by radiotherapy or radiotherapy followed by IPGDP regimen chemotherapy. IPGDP regimen for both arms are 3 cycles. And the chemotherapy is repeated every 3 weeks..

The second part: recruiting extensive stage II ,stage III-IV, relapsed or refractory ENKL patients. Patients receive 6 cycles of IPGDP regimen chemotherapy. And the chemotherapy is repeated every 3 weeks.

DETAILED DESCRIPTION:
The first Part: Patients in IPGDP regimen chemotherapy followed by radiotherapy arm receive 3 cycles of IPGDP (ifosfamide 1.2g/m2 iv on days 3-5; pegaspargase 2000U/m2 im on day 1; gemcitabine 800mg/m2 iv on days 3,8; cisplatin 25 mg/m2 iv on days 3-5; dexamethasone 20mg/m2 iv on days 3-6) chemotherapy. Then patients undergo radiotherapy. If the disease is considered to progress or as stable during chemotherapy, the patient will directly receive radiotherapy. Patients in another arm receive radiotherapy followed by IPGDP regimen chemotherapy. IPGDP regimen for both arms are 3 cycles, which is repeated every 3 weeks.

The second Part: Patients receive 6 cycles of ifosfamide 1.2g/m2 iv on days 3-5; pegaspargase 2000U/m2 im on day 1; gemcitabine 800mg/m2 iv on days 3,8; cisplatin 25 mg/m2 iv on days 3-5; dexamethasone 20mg/m2 iv on days 3-6. IPGDP regimen is repeated every 3 weeks. If the disease is considered to progress or as stable after 2 cycles or 4 cycles of chemotherapy, the patient will withdraw from this study.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of Extranodal Natural Killer/T-Cell Lymphoma, Nasal Type(ENKL)
* untreated ENKL patients of extensive stage I and limited stage II ( only referring to patients with the invasion of Waldeyer's ring and neck lymph node) confirmed by imaging examination; extensive stage II ,stage III-IV, relapsed or refractory ENKL patients confirmed by imaging examination
* age 18-65 years
* at least one measurable lesions
* Eastern Cooperative Oncology Group (ECOG) of 0 to 1
* a life expectancy of at least 12 weeks
* Adequate organ function including the following:

Bone marrow: absolute neutrophil count (ANC) >or equal to 1.5 * 109/L, platelets >or equal to 100 *109/L, hemoglobin > or equal to 9g/dL.

Hepatic: bilirubin < or equal to 2 x ULN; aspartate transaminase (AST) and alanine transaminase (ALT) < or equal to 2.5 x ULN (AST, ALT < or equal to 5 x ULN is acceptable if liver has been involved).

Renal: serum creatinine < or equal to 1.5 x ULN. Coagulation function :activated partial thromboplastin time < or equal to 1.5 x ULN, fibrinogen > or equal to 0.75 times of the lower limit of the normal value, INR < or equal to 1.5 x ULN.

* informed consent signed by patients prior to commencement of the study
* pregnancy test of Women of childbearing must be negative at the beginning of 7 days before treatment; surgical sterilization or taking contraceptive measures during treatment and three months after the end of treatment for males.

Exclusion Criteria:

* severe allergies to the investigational drugs
* patients who had received unauthorized drugs or drugs of other trials within 4 weeks prior to the study
* Severe or unstable systemic disease，serious neurological or psychiatric diseases including seizures or dementia
* organ function including the following: Bone marrow: absolute neutrophil count (ANC) < 1.5 * 109/L, platelets<100 *109/L, hemoglobin < 9g/dL.

Hepatic: bilirubin > 2 x ULN; aspartate transaminase (AST) and alanine transaminase (ALT) >2.5 x ULN (AST, ALT > 5 x ULN is acceptable if liver has been involved).

Renal: serum creatinine > 1.5 x ULN. Abnormal Coagulation function : such as activated partial thromboplastin time prolonged > 1.5 x ULN, fibrinogen < 0.75 times of the lower limit of the normal value, increased INR > 1.5 x ULN any other important clinical or laboratory abnormalities that are not appropriate for research

* Patients who had previously received treatment of this study, or withdrew from the study
* receiving any other anti-tumor therapy at the same time
* pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-09; Primary Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Institute/Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing
  - People's Hospital of Guangxi, Nanning
  - Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shanxi Dayi Hospital, Taiyuan
  - Shanxi Province Cancer Hospital, Taiyuan